CLINICAL TRIAL: NCT03622762
Title: Effect of the Administration of Green Tea Extract on Soluble RAGE and Kidney Disease in Patients With Diabetes Mellitus Type 2
Brief Title: Green Tea Extract on Soluble RAGE in Patients With Diabetic Nephropathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Fernando Grover Paez, Investigador Principal, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUCS-INTEC-MV-ERVE-06
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Diabetic Nephropathy Type 2
Keywords: Green tea extract; Kidney damage; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tea; Sunphenon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green tea extract (Experimental): In male and female population, with a diagnosis of Diabetes Mellitus type 2, under treatment with hypoglycemic agents and / or insulin and kidney damage grade 2 - 3a according to classification of the KDIGO guidelines
  Interventions: Drug: green tea extract
- Placebo (Placebo Comparator): In male and female population, with a diagnosis of Diabetes Mellitus type 2, under treatment with hypoglycemic agents and / or insulin and kidney damage grade 2 - 3a according to classification of the KDIGO guidelines
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: green tea extract — Capsules of green tea extract, 400 mg twice a day, fasting
  Other Names: Sunphenon
  Arms: Green tea extract
Drug: Placebo — Placebo capsules, 400 mg twice daily fasting
  Other Names: Calcined magnesium
  Arms: Placebo

SUMMARY:
Diabetic nephropathy is one of the most feared complications of Diabetes Mellitus type 2, characterized mainly by the decrease in the glomerular filtration rate and an increase in protein secretion by the kidney, that results in proteinuria. This has led to the development of intensive treatment regimens for patients with diabetes and preventive measures since once the complications have already presented the improvement of glycemic control alone may not be enough, to prevent the progression of pathological processes. Currently, interventions to delay the progression of kidney damage, include changes in lifestyle, nutritional advice and regular exercise, achieve optimal levels in glycemic control and use of pharmacological therapies with nephroprotector, angiotensin II receptor blocker (ARBs) and angiotensin-converting enzyme inhibitors (ACEIs). The most important biochemical mechanism proposed for this progression is the excessive binding of glucose to proteins, better described as the final products of advanced glycosylation (AGEs); the interaction of AGEs with its receptor (RAGE), participates in the metabolic and biochemical pathways in intracellular signaling, either by favoring or aggravating cell nephron damage. Recently, numerous RAGE isoforms have been described as: soluble RAGE, which are devoid of cytoplasmic domains, which bind to ligands that include AGEs and can antagonize intracellular signaling. Therefore, the need to seek for alternative therapies like nutraceuticals is arising, mainly due to its low toxicity and lower cost. Such is the case of green tea extract, which due to its chemical composition, especially of flavonoids that generate antioxidant and anti-inflammatory effects, In vivo and in clinical trials have shown that it could impact the progression of the diabetic neuropathy , through the modulation of the biological process, including molecular and biochemical pathways such as release of soluble RAGE.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the effect of the administration of green tea extract on soluble RAGE and renal damage in patients with Type 2 Diabetes Mellitus, by means of a clinical trial, double blind, with randomization and placebo control group. In male and female population, with a diagnosis of Diabetes Mellitus type 2, under treatment with hypoglycemic agents and / or insulin and kidney damage, 2 - 3a grade according to classification of the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines and HbA1c levels 9 - 12% who sign the letter of consent under information, from 35 to 65 years of age, residents of the metropolitan area of Guadalajara.

All patients who meet the selection criteria and who sign their informed consent will be given the clinical history, as well as anthropometric and laboratory determinations. Once these values are known, the intervention will proceed with the research product, extract of green tea 400 mg twice a day or placebo 400 mg twice a day, this will be according to the technique of masking by the closed envelope technique for 12 weeks. Patients will be evaluated at 30, 60 and 90 days of intervention, for attachment assessment, tolerability of treatment, side effects and laboratory safety determinations. At the end of the 12 weeks of the intervention, the anthropometric and laboratory determinations will be made again as well as the determination of soluble RAGE by means of Elisa sandwich type, in serum obtained at the beginning and at 12 weeks of intervention.

The database will be developed in the statistical program Statistical software (SPSS) version 21.0. The qualitative variables will be expressed in frequencies and percentages, while the quantitative variables will be expressed in means and standard deviations, the normality test will be carried out through the Kolmogorov-Smirnov test and, according to the result, it will be decided for the analysis intra group perform paired t or Wilcoxon method and for intergroup t student or Mann-Whitney U. A value of p ≤0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* People of both sexes
* Age from 40 to 65 years
* Signature of consent under information
* Diagnosis of type 2 diabetes mellituswith stable pharmacological treatment
* Glomerular filtration rate between 89 - 45 ml / min / 1.73 m2
* Albumin / creatinine ratio ≤ 30 - 300 mg / min
* HbA1c levels 7 - 12%
* Body mass index - 34.9

Exclusion Criteria:

* Glomerular filtration rat lower than 44 ml / min / 1.73 m2
* Albumin / creatinine ratio ≥ 300
* Other causes of kidney disease
* Other types of Diabetes
* Liver, thyroid or heart diseases
* Intolerance related to green tea or placebo components
* Use of antioxidant supplements
* Active alcoholism
* Patients with pregnancy or without a safe contraceptive method
* Patients in breastfeeding period

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-03-15 (Estimated); Study Completion 2019-06-20 (Estimated)

PRIMARY OUTCOMES:
Soluble RAGE concentration | 90 days
  Before and after the intervention using the serum extracted from the patient using sandwich ELISA.

SECONDARY OUTCOMES:
Glomerular filtration rate | 90 days
  Before and after the intervention, it will be evaluated by means of a determination of serum creatinine, which will be analyzed with the spectrophotometry method and from its result the glomerular filtration rate is calculated.
Albumin/creatinine ratio | 90 days
  Before and after intervention by spectrophotometry
Fasting plasma glucose | 90 days
  Before and after intervention spectrophotometry
Glycated Hemoglobin concentration | 90 days
  It will be analyzed by liquid chromatography
Systolic and diastolic arterial pressure | 90 days
  Before and after intervention using a digital baumanometer
Alanine aminotransferase | 90 days
  Before and after intervention by spectrophotometry
Aspartate aminotransferase | 90 days
  Before and after intervention by spectrophotometry

OTHER OUTCOMES:
Total cholesterol | 90 days
  Before and after intervention by spectrophotometry
triglycerides | 90 days
  Before and after intervention by spectrophotometry
High-density lipoprotein cholesterol | 90 days
  Before and after intervention by spectrophotometry
Low-density lipoprotein cholesterol | 90 days
  Before and after intervention by friedewall formula
Weight and visceral fat % | 90 days
  Before and after intervention using a vascula of impedance

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barocio-Pantoja M, Quezada-Fernandez P, Cardona-Muller D, Jimenez-Cazarez MB, Larios-Cardenas M, Gonzalez-Radillo OI, Garcia-Sanchez A, Carmona-Huerta J, Chavez-Guzman AN, Diaz-Preciado PA, Balleza-Alejandri R, Pascoe-Gonzalez S, Grover-Paez F. Green Tea Extract Increases Soluble RAGE and Improves Renal Function in Patients with Diabetic Nephropathy. J Med Food. 2021 Dec;24(12):1264-1270. doi: 10.1089/jmf.2020.0212. Epub 2021 Nov 17. PMID 34788550